# Statistical analysis plan Protocol 350A

### Trial NCT02475070

Study of the Effect of Vildagliptin versus Dapagliflozin on Glucagon

Response to Mixed Meal in Metformin-treated Subjects with Type 2

### **Diabetes**

#### Glucagon

Comparison between the two groups are performed with parametric t-test for glucagon in samples taken at -5, 15, 30, 45, 60, 90, 120, 180 and 240 min after meal ingestion and area under the 240 min curve (AUC) for glucagon

## Insulin, C-peptide, GIP and GLP-1

Comparison between the two groups are performed with parametric t-test for insulin, C-peptide, intact and total GIP and GLP-1 samples taken at -5, 15, 30, 45, 60, 90, 120, 180 and 240 min after meal ingestion and area under the 240 min curve (AUC) for insulin, C-peptide, intact and total GIP and GLP-1.

Lund, March 28, 2016

Bo Ahrén, PI